CLINICAL TRIAL: NCT00356954
Title: N-Acetylcysteine vs. Ascorbic Acid for Prevention of Contrast Induced Nephropathy in Renal Insufficiency Undergoing Coronary Catheterization: NASPI Study-A Randomized Controlled Trial
Brief Title: NASPI: N-Acetylcysteine vs. Ascorbic Acid for Prevention of Contrast Induced Nephropathy in Renal Insufficiency Undergoing Coronary Catheterization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-0509-517-158-2
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2006-11-27 (Estimated); Status verified 2006-11

CONDITIONS: Kidney Failure
Keywords: Kidney failure; Contrast media; Antioxidant; Prevention
MeSH Terms: conditions — Renal Insufficiency | interventions — Ascorbic Acid

INTERVENTIONS:
Drug: N-acetylcystein
Drug: ascorbic acid

SUMMARY:
The contrast induced nephropathy (CIN) has been known to be associated with significant clinical and economic consequences. Many studies were performed to find the pathophysiology and preventive measures for CIN. But the results were somewhat frustrating. Recently, it has been reported that the N-acetylcysteine and ascorbic acid might have preventive effects for CIN by their antioxidant effects.There have been no study to compare these two antioxidant.

DETAILED DESCRIPTION:
N-acetylcysteine and ascorbic acid may prevent the CIN in the patients with underlying renal insufficiency who is undergoing the coronary angiography. The effect may derive from the antioxidant function of these two antioxidant. We studied to find which of the two antioxidants is more beneficial in prevention of CIN

ELIGIBILITY:
Inclusion Criteria:

* Stable Angina pectoris patients
* Patients who required the coronary catheterization
* Creatinine clearance rates =<60 mL/min using the Cockcroft-Gault formula
* Age of 19 or over 19

Exclusion Criteria:

* Pregnancy
* Lactation
* Having received contrast media within 7 days of study entry
* Emergent coronary angiography
* Acute renal failure
* End-stage renal disease requiring dialysis
* History of hypersensitivity reaction to contrast media
* Cardiogenic shock
* Pulmonary edema
* Multiple myeloma
* Mechanical ventilation
* Parenteral use of diuretics
* Recent use of N-acetylcysteine
* Recent use of Ascorbic acid
* Recent use of statin
* Use of metformin or nonsteroidal anti-inflammatory drugs within 48 hours of the procedure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2005-02; Study Completion 2006-04

PRIMARY OUTCOMES:
The mean peak increase of serum creatinine concentration during day1 and day2.

SECONDARY OUTCOMES:
Incidence of contrast induced nephropathy, defined as either a relative increase in serum creatinine
from baseline of >=25% or an absolute increase of >=0.5mg/dL(44.2µmol/L) during days 1 and 2.
Proportion of patients exhibiting an increase in serum creatinine of >=0.5mg/dL(44.2µmol/L)
proportion with a >=1.0 mg/dL(88.4µmol/L) increase in serum creatinine;

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Ho Jo, M.D., Principal Investigator — Seoul National University Hospital, Department of Internal Medicine/ Cardiovascular Center, Hallym University Sacred Heart Hospital; Bon-Kwon Koo, M.D., Ph.D., Principal Investigator — Seoul National University Hospital, Department of Internal Medicine/ Cardiovascular Center; Hyo-Soo Kim, M.D.,Ph.D., Study Director — Seoul National University Hospital, Department of Internal Medicine/ Cardiovascular Center; Byung-Hee Oh, M.D., Ph.D., Study Chair — Seoul National University Hospital, Department of Internal Medicine/ Cardiovascular Center
Locations (1):
- Seoul National University Hospital , Cardiovascular Center, Seoul, South Korea